CLINICAL TRIAL: NCT01836575
Title: Phase III Trial of Single-Agent Pemetrexed (Alimta®) Versus the Combination of Carboplatin and Pemetrexed in Patients With Advanced Non-small-cell Lung Cancer and Performance Status of 2
Brief Title: Alimta® Versus Its Combination With Carboplatin in Advanced Non-small-cell Lung Cancer in Patients Performance Status 2
Acronym: PS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H3E-BL-O027-PS2; H3E - US -I023 (Other: INCA-Lung001); INCA-Lung001 (Other: INCA - Brazilian National Cancer Institute)
Record Dates: First submitted 2010-12-30; First posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Advanced NSCLC; PS2; Pemetrexed; First line; non squamous
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Glucose; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B (Experimental): Pemetrexed, 500mg/m2 + appropriate vitamin supplementation + Carboplatin [Target AUC 5 IV infusion,based on Calvert formula,GFR estimated using estimated creatinine clearance per Cockcroft and Gault formula, obtained prior to each cycle] + Antiemetic therapy at investigator's discretion.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin
- Arm A: (Active Comparator): Pemetrexed, 500mg/m2 + appropriate vitamin supplementation + Antiemetic therapy at investigator's discretion.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed, 500 mg/m2 + Pretreatment [dexamethasone + vitamin B12 + folic acid, as per pemetrexed label] + Antiemetic therapy at investigator's discretion.
  Other Names: Arm A - active comparator Pemetrexed (Alimta).
Drug: Carboplatin — Carboplatin [Target AUC 5 IV infusion,based on Calvert formula,GFR estimated using estimated creatinine clearance per Cockcroft and Gault formula, obtained prior to each cycle].
  Other Names: Carboplatin AUC 5 IV in 5% dextrose or 0.9% sodium chloride.
  Arms: Arm B

SUMMARY:
Optimal management of patients with advanced NSCLC and with PS 2 remains controversial and underrepresented in clinical trials, typically accounting for 5 to 10% of enrolled patients. Patient PS 2 proportion in population-based studies is considerably higher than that included in clinical trials. Management of patients with PS of 2 in clinical practice is empirical and inconsistent. Patients have median overall survival of 3 to 5 months in randomized trials, and treatment options include best supportive care, single-agent and combination chemotherapy. Retrospective studies have suggested that patients PS 2 may benefit from first-line chemotherapy in terms of symptom improvement and overall survival. In many of these studies, single-agent chemotherapy was compared with best supportive care alone. Data on the role of cisplatin-based combinations for patients with PS 2 is more scant, with one study questioning its benefit, and another interrupting accrual because of undue toxicity. With regards to carboplatin, the Cancer and Leukemia Group B (CALGB) study 9730 compared paclitaxel plus carboplatin versus paclitaxel alone in a subgroup of 107 patients with PS 2; the median overall survival was significantly longer in group treated with combination chemotherapy (4.7 versus 2.4 months). Combination chemotherapy with carboplatin and paclitaxel also produced a statistically significantly higher incidence of severe hematological and non-hematological toxicities. On the basis of aforementioned results, a recent European panel stated that carboplatin-based or low-dose cisplatin-based doublets might represent alternative options to single-agent chemoterapy in patients PS 2. Outside clinical trials, single-agent chemotherapy with a 3rd generation agent remains valid option for patients PS2. Results demonstrate that pemetrexed is an agent with established single-agent activity in NSCLC, and suggest it is a potential candidate for combinations with platinum and other agents currently utilized for patients with advanced NSCLC. Favorable toxicity profile of pemetrexed suggests that this agent is an ideal candidate for single agent testing and in combination among patients with PS 2. Substantial doubt remains in the comparative benefit from monotherapy versus combination. Starting dose and schedule of pemetrexed were set for this study based on its current labeling in the 2nd line treatment of metastatic NSCLC and 1st line treatment of malignant pleural mesothelioma.

DETAILED DESCRIPTION:
This is a Phase III, open label, randomized study to enroll 228 patients with advanced in a 1:1 ratio at the time of registration. Patients in Arm A will receive pemetrexed, 500 mg/m2, with appropriate vitamin supplementation; patients in Arm B will receive the same dose and schedule of pemetrexed as in Arm A, in combination with carboplatin, AUC of 5. For the purpose of the study, treatment (Arm A or Arm B) will consist of up to four cycles of therapy (repeated every 21 days). Primary endpoint of the study is overall survival; secondary endpoints include toxicity, response rate, and progression-free survival. At the time of analysis, patients will be stratified according to age (≥ 70 versus < 70 years), disease stage (IIIB versus IV), site, and weight loss (≥ 5 Kg versus < 5 Kg).

The dose of carboplatin will be determined according to the formula developed by Calvert et al., which is shown in equation [1] below and uses the estimated creatinine clearance according to the method of Cockcroft and Gault for estimation of the glomerular filtration rate (GFR) (equation [2] below):

1. Dose of carboplatin (mg) = Target AUC x (GFR + 25)
2. GFR = (140 - Age) x Weight/(72 x serum creatinine) (multiply by 0.85 in women) Sample Size and Expected Accrual In the CALGB 9730 study of advanced NSCLC, first-line treatment with paclitaxel plus carboplatin resulted in a median overall survival of 4.7 months among patients with a performance status of 2. In the ECOG 1594 study, the median overall survival of patients with a performance status of 2 who were treated with platinum-based doublets was 4.1 months. Approximately 208 eligible patients are needed to provide 80% power to detect a difference between the two treatment arms with a two-sided type I error of 0.05, assuming that pemetrexed plus carboplatin will result in a median survival of at least 4.3 months, and pemetrexed alone 2.9 months. An additional 20 patients will be accrued to account for an early dropout rate of 10%, for a total of 228 patients. It is anticipated that the accrual time will be approximately 22 months and patients will be followed for 1 year after completion of treatment; therefore, 2 years and 10 months will be needed to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed NSCLC in stage IIIB (with a cytologically positive pleural or pericardial effusion) or stage IV, according to the sixth edition of the American Joint Committee on Cancer (AJCC) Cancer Staging Manual37;
* Age > 18 years;
* No prior chemotherapy, including adjuvant or neoadjuvant therapy, for the treatment of NSCLC;
* Histological confirmation of any non-squamous histological type of NSCLC, given the recent findings of treatment benefit in this population44;
* ECOG performance status of 2;
* At least 3 weeks must have elapsed since major surgery, and at least 1 week since mediastinoscopy, pleuroscopy, or thoracostomy;
* Patients must have measurable disease, defined as lesions that can be accurately measured in at least 1 dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques (computed tomography [CT] or magnetic resonance imaging [MRI] scan) or as ≥ 10 mm with spiral CT scan;
* Adequate organ function as indicated by the following:

  * White blood cell (WBC) count ≥ 3500/mm3
  * Absolute neutrophil count (ANC) ≥1500/mm3
  * Hemoglobin ≥ 9.0 g/dL
  * Platelet count ≥ 100,000/ mm3
  * Total bilirubin ≤ 2 times the upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the ULN, unless liver metastases present, in which case AST and ALT have to be ≤ 5 times the ULN
  * Estimated glomerular filtration rate (GFR) ≥ 45 mL/min
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration;
* Fertile patients (male or female) must agree to use an acceptable method of contraception to avoid pregnancy for the duration of the study and for 3 months thereafter;
* Patients must sign an Informed Consent Form;
* Have the ability to take folic acid, Vitamin B12, and dexamethasone according to protocol requirements;

Exclusion Criteria:

* ECOG performance status other than 2;
* Prior chemotherapy for the treatment of NSCLC;
* Lesions that have been irradiated cannot be included as sites of measurable disease. If the only measurable lesion was previously irradiated the patient cannot be included;
* Symptomatic central nervous system (CNS) metastases. Prior CNS metastases are allowed if the patient is neurologically stable and not receiving corticosteroids;
* Serious uncontrolled intercurrent medical or psychiatric illness;
* Active and ongoing systemic infection;
* Second primary malignancy (except in situ carcinoma of the cervix, in situ carcinoma of the bladder, adequately treated basal-cell carcinoma of the skin, adequately treated squamous-cell carcinoma of the skin, T1 vocal cord cancer in remission, or prior malignancy treated more than 5 years prior to enrollment and without recurrence);
* Known hypersensitivity to pemetrexed;
* known hypersensitivity to carboplatin;
* Pregnancy or lactation;
* Use of any investigational agent within 30 days prior to enrollment into the study;
* Unable to discontinue administration of non-steroidal anti-inflammatory (NSAIDSs) agents for 2 days before, the day of and 2 days after the dose of pemetrexed, in the case of NSAIDs with short half-life, such as ibuprofen (total of 5 days), in patients with a GFR between 45 and 79 mL/min; and for 5 days before, the day of and 2 days after the dose of pemetrexed, in the case of NSAIDs with long half-life (total of 8 days, see 7.4.2) in all patients; patients with a GFR ≥ 80 mL/min may receive concomitant study treatment and ibuprofen or aspirin (≤ 1.3 g/day);
* Inability to comply with requirements and procedures of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2008-04; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | From ICF signature date until e until death date for any cause
  Each patient will be followed from inclusion date in the study (ICF signature) until the death date for any cause, whichever came first, assessed up to one year after completion of study treatment. Primary objective of this study is to determine and compare the overall survival produced by pemetrexed as a single-agent and by the combination of pemetrexed plus carboplatin in a patient with previously untreated, advanced non-squamous NSCLC and an ECOG Performance status of 2.

SECONDARY OUTCOMES:
Safety evaluation | Serious Adverse Event every 6 months
  Planned interim analysis for the 46 death events, and cut off for patients at V3 to V6, every 06 months as average. Patients with at least any study treatment dose were included in safety analyses, focused on toxicity grades 3-4. Toxicity evaluation from date of last treatment dose until 1 month of follow up visit date, and every cycle according CTCAE v3.0 for study dose adjustment as per guidelines based on episodes of febrile neutropenia; grade 4 thrombocytopenia and/or bleeding; and any grade 3 or 4 non-hematologic toxicity except nausea/emesis. Safety evaluation for medical conditions, symptoms or signs, laboratory parameters as per protocol criteria, disregarding disease progression when unrelated drugs or any procedure of study.
Progression free survival | Final data analysis: Sep/2012
  Progression free survival evaluated by RECIST criteria, as described in protocol. Time for Progression free survival will be measured from date of first treatment dose to either date a patient is first recorded as disease progression (even for a withdrawn patient due to toxicity), or the date of death due to any causes before progression. Patient lost of follow up will be censored from the last contact date. Patients starting new treatment before disease progression will be censored at that date of starting new treatment. A patient who dies without disease progression the time for this assessment will be last follow-up date.
Response Rate | Final data analysis: Sep/2012
  Objective response rate evaluated by RECIST criteria as described in protocol. From those patients with tumoral response, the duration of response is measured from the date of first response evidence (Complete and Partial Responses) until first recorded as disease progression, or date of death to any causes before progression. Duration for tumoral response will be censored in the last follow up date for those patients with tumoral response who still alive and has not progressed.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos G Ferreira, PhD, Principal Investigator — National Cancer Institute, France; Rogerio Lilenbaum, MD, Principal Investigator — The Mount Sinai Comprehensive Cancer Center; Carlos Henrique E Barrios, MD, Principal Investigator — Pontifícia Universidade Católica do RS; Carlos Augusto M. Beato, MD, Principal Investigator — Hospital Amaral Carvalho; José Rodrigues, MD, Principal Investigator — Instituto do Câncer Arnaldo Vieira Carvalho - ICAVC; Yeni Neron, MD, Principal Investigator — Centro de Pesquisas Oncológicas - CEPON; André Murad, PhD, Principal Investigator — Lifecenter Hospital; Ronaldo A Ribeiro, PhD, Principal Investigator — Instituto do Câncer do Ceará - ICC; Fábio Franke, MD, Principal Investigator — Hospital de Caridade de Ijuí - CACON; Mauro Zukin, MD, Principal Investigator — National Cancer Institute, France
Locations (9):
- The Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida, United States
- Brazil (8):
  - Instituto do Câncer do Ceará - ICC, Fortaleza, Ceará
  - Hospital Lifecenter, Belo Horizonte, Minas Gerais
  - INCA, Rio de Janeiro, Rio de Janeiro
  - Hospital Caridade de Ijuí - CACON, Ijuí, Rio Grande do Sul
  - Hospital São Lucas, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncológicas - CEPON, Florianópolis, Santa Catarina
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto do Câncer Arnaldo Vieira de Carvalho, São Paulo, São Paulo

REFERENCES:
- [Derived] Gijtenbeek RG, de Jong K, Venmans BJ, van Vollenhoven FH, Ten Brinke A, Van der Wekken AJ, van Geffen WH. Best first-line therapy for people with advanced non-small cell lung cancer, performance status 2 without a targetable mutation or with an unknown mutation status. Cochrane Database Syst Rev. 2023 Jul 7;7(7):CD013382. doi: 10.1002/14651858.CD013382.pub2. PMID 37419867
- [Derived] Zukin M, Barrios CH, Pereira JR, Ribeiro Rde A, Beato CA, do Nascimento YN, Murad A, Franke FA, Precivale M, Araujo LH, Baldotto CS, Vieira FM, Small IA, Ferreira CG, Lilenbaum RC. Randomized phase III trial of single-agent pemetrexed versus carboplatin and pemetrexed in patients with advanced non-small-cell lung cancer and Eastern Cooperative Oncology Group performance status of 2. J Clin Oncol. 2013 Aug 10;31(23):2849-53. doi: 10.1200/JCO.2012.48.1911. Epub 2013 Jun 17. PMID 23775961